CLINICAL TRIAL: NCT05597787
Title: Implementing Stigma Reduction Tools Via a Popular Teletraining Platform to Reduce Clinician Stigma and Disparities in HIV Testing, Prevention, and Linkage to Care in Malaysia
Brief Title: HIV-Related Stigma Intervention for Malaysian Clinicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: R34MH124390 (NIH)
Record Dates: First submitted 2022-07-25; First posted 2022-10-28 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-01

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIV Connect (Active Comparator): Participants randomized to this condition will complete HIV Connect, which is an online course developed by the Malaysian Society of HIV Medicine designed to educate primary care physicians in Malaysia about HIV. It consists of a series of modules featuring HIV infectious disease experts who instruct on topics including epidemiology and natural history of HIV, pre-exposure prophylaxis (PrEP) and post-exposure prophylaxis (PEP), sexual history taking and STI testing, and others.
  Interventions: Behavioral: HIV Connect
- Project ECHO for HIV Prevention (Active Comparator): Participants randomized to this condition will receive Project ECHO for HIV Prevention, without added evidence-based stigma reduction tools. Participants will meet with the Project ECHO Hub specialists and their learning community on a bi-weekly basis for 60 minutes over the course of 9 months. Each session will feature a didactic training incorporating standardized procedures for HIV testing, prevention, and/or linkage to care, and patient-case presentation and discussion.
  Interventions: Behavioral: Project ECHO for HIV Prevention
- Project ECHO for HIV Prevention + Stigma Reduction (Experimental): Participants randomized to this condition will receive the Project ECHO for HIV Prevention intervention with added evidence-based stigma reduction tools. Participants will meet with the Project ECHO Hub specialists and their learning community on a bi-weekly basis for 60 minutes over the course of 9 months. Each session will feature a didactic training incorporating standardized procedures for HIV testing, prevention, and/or linkage to care, and patient-case presentation and discussion.
  Interventions: Behavioral: Project ECHO for HIV Prevention and Stigma Reduction

INTERVENTIONS:
Behavioral: HIV Connect — online education and clinical skills
  Arms: HIV Connect
Behavioral: Project ECHO for HIV Prevention — education and clinical skills
  Arms: Project ECHO for HIV Prevention
Behavioral: Project ECHO for HIV Prevention and Stigma Reduction — education, clinical skills and contact
  Arms: Project ECHO for HIV Prevention + Stigma Reduction

SUMMARY:
Key populations at risk of HIV (including men who have sex with men, people who inject drugs, transgender women, and female sex workers) are more likely to be infected with HIV but less likely than members of the general population to know of their HIV status, receive HIV prevention counseling, or be linked to HIV care services. Clinician stigma towards these groups remains a potent and persistent driver of these HIV disparities in many places of the world. The investigators propose to incorporate evidence-based stigma reduction tools into a popular teletraining platform for clinicians and pilot test the resulting intervention (Project ECHO® for HIV Prevention and Stigma Reduction) with clinicians in Malaysia, a context wherein clinician stigma and HIV disparities are substantial.

ELIGIBILITY:
Inclusion Criteria:

* practicing general practitioner or family medicine specialist in Malaysia

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Because of the risks and sensitivities of this study, only completely de-identified data will be shared under a use agreement. Data-sharing agreements must provide for: (1) a commitment to using the data only for research purposes, (2) a commitment to securing the data using appropriate computer technology and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Earnshaw VA, Collier ZK, Wong PL, Saifi R, Chong N, Ng RX, Azwa I, Basri S, Hassan ABA, Mousavi M, Omar SFS, Walters S, Haddad MS, Kamarulzaman A, Altice FL. Pilot randomized controlled trial to reduce HIV-related stigma among clinicians in Malaysia via project ECHO(R). AIDS Care. 2025 Aug;37(8):1313-1331. doi: 10.1080/09540121.2025.2534539. Epub 2025 Jul 30. PMID 40736373
- [Derived] Chong N, Azwa I, Hassan AA, Mousavi M, Wong PL, Ng RX, Saifi R, Basri S, Omar SFS, Walters SM, Collier ZK, Haddad MS, Altice FL, Kamarulzaman A, Earnshaw VA. Strengthening HIV Activism Among Clinicians in Malaysia: A Randomised Controlled Trial. AIDS Behav. 2025 Dec;29(12):3931-3939. doi: 10.1007/s10461-025-04829-1. Epub 2025 Jul 21. PMID 40691430

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Advertisements were posted to Malaysian medical groups (i.e., Family Medicine Association, Malaysian Medicine Association, Malaysian Primary Care Network, Doctors Only Bulletin Board System) between May and July 2022.
Pre-assignment Details: n=411 individuals accessed the registration link. Of these, n=257 were excluded because they declined to participate in the study, were withdrawn because they provided incomplete registration data or their identity could not be verified, or were waitlisted. Of the remaining individuals, n=26 were allocated to an intervention condition. Individuals who did not receive an intervention withdrew, became non-responsive to communication from the project coordinator, or were waitlisted.
Period: Overall Study
Arm/Group | HIV Connect | Project ECHO for HIV Prevention | Project ECHO for HIV Prevention + Stigma Reduction
Started | 26 | 26 | 26
Completed | 26 | 26 | 25
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The participant who withdrew from the Project ECHO for HIV Prevention and Stigma Reduction condition completed follow-up surveys, and so is included in analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Connect | Project ECHO for HIV Prevention | Project ECHO for HIV Prevention + Stigma Reduction | Total
Number analyzed (Participants) | 26 | 26 | 26 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.42 (6.37) | 36.50 (4.05) | 38.23 (7.28) | 37.38 (6.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 10 | 32
  Male | 13 | 17 | 16 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Malay | 4 | 14 | 10 | 28
  Chinese | 16 | 6 | 13 | 35
  Indian | 5 | 6 | 13 | 24
  Other | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Malaysia | 26 | 26 | 26 | 78

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention
Description: Measured with Acceptability of Intervention Measure. Theoretical or possible range of scores is 1-5, and actual range was 3.50-5. Higher scores indicate greater acceptability.
Time Frame: Month 9 Assessment
Population: Two participants in the Project ECHO for HIV Prevention Condition did not complete the month 9 survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIV Connect | Project ECHO for HIV Prevention | Project ECHO for HIV Prevention + Stigma Reduction
Number analyzed (Participants) | 26 | 24 | 26
score on a scale | 4.22 (0.44) | 4.72 (0.39) | 4.45 (0.48)

2. Primary Outcome: Feasibility of Intervention
Description: Measured with Feasibility of Intervention Measure. Theoretical or possible range of scores is 1-5, and actual range was 3.25-5. Higher scores indicate greater feasibility.
Time Frame: Month 9 Assessment
Population: Two participants in the Project ECHO for HIV Prevention Condition did not complete the final survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIV Connect | Project ECHO for HIV Prevention | Project ECHO for HIV Prevention + Stigma Reduction
Number analyzed (Participants) | 26 | 24 | 26
score on a scale | 4.22 (0.44) | 4.62 (0.45) | 4.32 (0.60)

3. Primary Outcome: Stigma Reduction: Prejudice
Description: Measured with Feelings Thermometers. Positive/Negative affect is measured on 0-100 point scale, with higher scores indicating more prejudice.
Time Frame: Month 9 Assessment
Population: Two participants in the Project ECHO for HIV Prevention condition did not complete the final survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIV Connect | Project ECHO for HIV Prevention | Project ECHO for HIV Prevention + Stigma Reduction
Number analyzed (Participants) | 26 | 24 | 26
score on a scale | 29.13 (18.84) | 23.28 (20.50) | 32.07 (15.36)

4. Primary Outcome: Stigma Reduction: Stereotypes
Description: Measured with subscale of Multidimensional HIV-Related Stigma Scale. Theoretical or possible range of scores is 1-5, and actual range was 1-3.44. Higher scores indicate greater stereotypes.
Time Frame: Month 9 Assessment
Population: Two participants in the Project ECHO for HIV Prevention condition did not complete the final survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIV Connect | Project ECHO for HIV Prevention | Project ECHO for HIV Prevention + Stigma Reduction
Number analyzed (Participants) | 26 | 24 | 26
score on a scale | 2.55 (0.50) | 2.01 (0.59) | 2.32 (0.69)

5. Primary Outcome: Stigma Reduction: Discrimination
Description: Measured with subscale of Multidimensional HIV-Related Stigma Scale. Theoretical or possible range of scores is 1-5, and actual range was 1-5. Higher scores indicate greater discrimination.
Time Frame: Month 9 Assessment
Population: Two participants in the Project ECHO for HIV Prevention condition did not complete the final survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIV Connect | Project ECHO for HIV Prevention | Project ECHO for HIV Prevention + Stigma Reduction
Number analyzed (Participants) | 26 | 24 | 26
score on a scale | 4.44 (0.50) | 4.67 (0.85) | 4.64 (0.42)

6. Secondary Outcome: HIV Prevention Procedures: HIV Testing
Description: Measured with weekly diary of HIV tests performed. Number of HIV tests will be summed over duration of intervention.
Time Frame: Cumulative over 9 month intervention
Population: Submission of procedures data was inconsistent, with many participants missing submissions in each condition.
Measure: Mean (Standard Deviation); unit: number of HIV tests
Arm/Group | HIV Connect | Project ECHO for HIV Prevention | Project ECHO for HIV Prevention + Stigma Reduction
Number analyzed (Participants) | 19 | 15 | 18
number of HIV tests | 21.54 (45.14) | 2.65 (6.17) | 10.46 (46.24)

7. Secondary Outcome: HIV Prevention Procedures: PrEP Prescriptions
Description: Measured with weekly diary of PrEP prescriptions. Number of PrEP prescriptions will be summed over duration of intervention.
Time Frame: Cumulative over 9 month intervention
Population: Submission of procedures data was inconsistent, with many participants missing submissions in each condition.
Measure: Mean (Standard Deviation); unit: number of PrEP prescriptions
Arm/Group | HIV Connect | Project ECHO for HIV Prevention | Project ECHO for HIV Prevention + Stigma Reduction
Number analyzed (Participants) | 19 | 15 | 18
number of PrEP prescriptions | 2.04 (8.80) | 0.07 (0.27) | 0.11 (0.43)

ADVERSE EVENTS:
Time Frame: 9 months
Description: The definition of adverse event and/or serious adverse event did not differ from the clinicaltrials.gov definitions for this study.
Arm/Group | HIV Connect | Project ECHO for HIV Prevention | Project ECHO for HIV Prevention + Stigma Reduction
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT05597787/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT05597787/ICF_001.pdf